CLINICAL TRIAL: NCT00539669
Title: TAX + Carboplatin or Cisplatin 1st Line Post-Surgery Ovarian
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XRP6976I_2502
Record Dates: First submitted 2007-10-03; First posted 2007-10-04 (Estimated); Last update posted 2007-10-04 (Estimated); Status verified 2007-10

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: Docetaxel

SUMMARY:
Evaluate response rate of Docetaxel in combination with Carboplatin or Cisplatin as first line chemotherapy in epithelial ovarian cancer. Assess the progression free survival, tolerance, duration of response and survival in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian carcinoma. Patients with peritoneal carcinomatosis are also eligible, without necessarily having histological proof of a primary source in the ovary, provided that the tumour is not mucin-secreting, and that there is no evidence of a primary fallopian tube cancer (see exclusion criteria).
* Female, aged 18 or over- FIGO stages Ic-IV with or without successful cytoreductive surgery at staging laparotomy. Stage Ic patients will be limited to those with malignant cells in ascitic fluid, peritoneal washings or with tumour on the surface of the ovary
* Patients with ruptured capsule as the only evidence of stage Ic will not be eligible for entry into the study.

Exclusion Criteria:

* ECOG performance status > 2
* Prior treatment with chemotherapy or radiotherapy.
* Patients with, pre-existing fluid retention such as pleural effusion, pericardial effusion and ascites are not excluded from the study, but should be monitored closely for any deterioration. Efforts should be made to determine by cytological analysis whether any significant pre-existing fluid collections are due to ovarian cancer, and subsequent drainage is recommended before initiating chemotherapy.
* Inadequate bone marrow function defined as neutrophils < 1.5 x 109/l or platelets < 100 x 109/l.
* Inadequate renal function as defined by serum creatinine > 1.25 x upper limit of normal.
* Inadequate liver function as defined by bilirubin > upper limit of normal or AST/ALT > 1.5 x upper limit of normal or ALP > 3 x upper limit of normal.
* Concurrent severe and/or uncontrolled co-morbid medical condition (i.e. uncontrolled infection, hypertension, ischaemic heart disease, myocardial infarction within previous 6 months, congestive heart failure)
* Patients with mixed mesodermal tumours.
* Patients with borderline ovarian tumours or tumours termed 'possibly malignant'.
* Adenocarcinoma of unknown origin, if histologically shown to be mucin-secreting cancer or thought to be possible primary fallopian tube carcinoma.
* History of previous malignancy within the previous 5 years (except curatively treated carcinoma in situ of the uterine cervix, or basal cell carcinoma of the skin), or concurrent malignancy (e.g. coexisting endometrial cancer) .
* History of prior serious allergic reactions (e.g. anaphylactic shock).
* History of other relative contraindications to corticosteroid administration
* Pregnant or lactating women (or potentially fertile women not using adequate contraception).
* Symptomatic peripheral neuropathy > NCIC-CTC grade II.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-03

PRIMARY OUTCOMES:
The response rate will be determined by the number of patients with complete and partial responses according to the Modified SWOG Response Criteria. The progression free survival, duration of response and survival are evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Hyang Rim Kim, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Seoul, South Korea